CLINICAL TRIAL: NCT07022756
Title: Personalized Outreach for Equitable Treatment in Rheumatology: A Randomized Controlled Trial of Patient Outreach and Honoraria in an Inner City Rheumatology Clinic
Brief Title: Personalized Outreach for Equitable Treatment in Rheumatology
Acronym: POET-Rheum
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Mary Pack Arthritis Center (Unknown)
Responsible Party: Principal Investigator, Alec Yu, Lead Investigator - Personalized Outreach for Equitable Treatment in Rheumatology, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: H24-03984
Record Dates: First submitted 2025-06-07; First posted 2025-06-15 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-07

CONDITIONS: Rheumatic Diseases; Inflammatory Arthritis; Rheumatoid Arthritis (RA); Psoriatic Arthritis (PsA); Connective Tissue Disease
Keywords: Rheumatology; Inflammatory Arthritis; Inner City Health
MeSH Terms: conditions — Rheumatic Diseases; Arthritis; Arthritis, Rheumatoid; Arthritis, Psoriatic; Connective Tissue Diseases | interventions — Community-Institutional Relations

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Honoraria Only (Active Comparator): Participants in this arm of the study will only receive honoraria and not outreach
  Interventions: Behavioral: Honoraria
- Honoraria and Outreach (Experimental): Participants in this arm of the study will receive both honoraria and outreach services
  Interventions: Behavioral: Honoraria; Behavioral: Outreach
- Historical Control (No Intervention): The attendance rate to follow-up appointments among all patients with inflammatory arthritis due to a rheumatic disease at the Pender Rheumatology Clinic from Jan 2023 to Jun 2025.

INTERVENTIONS:
Behavioral: Honoraria — A $20 honorarium for each appointment attended with completed bloodwork if requested.
  Arms: Honoraria Only; Honoraria and Outreach
Behavioral: Outreach — A personalized outreach service specific for rheumatic disease.
  Arms: Honoraria and Outreach

SUMMARY:
The primary goal of this study is to determine whether providing patient honoraria and/or outreach services can improve the attendance rate of appointments at an inner city rheumatology clinic in Vancouver, British Columbia.

The main question it aims to answer are:

* Does providing a financial honorarium ($20 for each follow-up appointment with completed bloodwork) improve attendance rate at an inner city rheumatology clinic?
* Does providing a personalized outreach service for rheumatic diseases improve attendance rate at an inner city rheumatology clinic?

The researchers will compare providing patient honoraria to providing both honoraria and outreach services, and compare each of these to the regular appointment schedule without honoraria or outreach.

Participants will:

* Undergo randomization to receive honoraria or honoraria and outreach services together
* Complete surveys about their health and understanding of their rheumatic disease at baseline, 3-month, and 6-month intervals
* Visit the clinic every month for check-ups and monitoring bloodwork if they are started on immunosuppressants for their condition

DETAILED DESCRIPTION:
Our study aims to enhance the existing twice-monthly rheumatology clinic at the Pender Community Health Centre with a rheumatology-specific outreach service for patients with inflammatory arthritis. This service will be provided by a rheumatology subspecialty trainee under the supervision of two attending rheumatologists. This will consist of biweekly phone calls, text messages, or home visits as per the patient's preference, at times flexible to patient needs. This will be in addition to monthly in-person assessment and bloodwork monitoring with adjustment as clinically indicated by their treating rheumatologist. Outreach services will include management of medications and side effects, proactive screening for infections, coordination of rheumatologic and general healthcare with their Primary Care Provider, social service navigation, and reminders for appointments and lab monitoring. All participants will be provided with a $20 honorarium for each in-person assessment they attend as part of the study.

The investigators will aim to enroll 20 participants between July 2025 and October 2025. Participants will be randomized to either honorarium with outreach or honorarium alone arms in a 1:1 fashion, stratified by housing status (unhoused and emergency sheltered in one strata, provisionally accommodated and stably housed in the second strata).

All enrolled participants will receive a $20 honorarium for each in-person assessment with completed monitoring bloodwork as requested by the treating rheumatologist. The program will last 6 months for each patient from time of enrolment, or until a patient chooses to leave the program, whichever is sooner. At baseline, participants will complete two surveys: one on their general health status, and one specific to their rheumatic disease. At the 3-month and 6-month visits, these surveys will be repeated, and a semi-structured interview will be completed to obtain feedback on the pilot program.

The outcomes of this study will inform how rheumatologists can better care for those who live with inflammatory arthritis and are also marginalized by extreme poverty and/or housing instability. The investigators plan on disseminating and discussing results with our participants, community members, inner city physicians, and rheumatologists. If there are specific positive themes or outcomes from the study, the investigators will advocate for additional resources to permit long-term implementation and further study to confirm results, make further improvements to our program, and improve generalizability.

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of inflammatory arthritis secondary to an autoimmune rheumatic disease
* Be attached to one of the Vancouver Coastal Health Community Health Centres for primary care
* Be willing to attend in-person appointments at Pender Community Health Centre
* Be at least 18 years of age and capable of consenting to participation
* Be able to receive medical care in English.

Exclusion Criteria:

* Have cognitive impairment or an untreated psychiatric condition that would severely impair ability to engage with outreach or treatment
* Have no reasonably reliable method of contact (phone, email, social media, etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-07-02 (Estimated); Primary Completion 2026-04 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Attendance at in-person follow-up appointments | Cumulative over 6 months
  Adherence to in-person follow-up measured by the ratio of appointments attended to appointments scheduled.

SECONDARY OUTCOMES:
Clinical Disease Activity Index (CDAI) | 3-month and 6-month intervals.
  The change in Clinical Disease Activity Index from baseline to 3-months and 6-months. The Clinical Disease Activity Index is a validated disease outcome measure in Inflammatory Arthritis ranging from 0 to 76. A higher score means a worse outcome.
Patient Qualitative Feedback | 3-month and 6-month intervals.
  Patient qualitative feedback on the program via semi-structured interview.
Patient Reported Understanding of Disease and Medications | 3-month and 6-month intervals.
  Patient Reported Understanding of Disease and Medications, as measured by likert scale at baseline, 3 months, and 6 months. The likert scale will range from 1 to 10, with higher scores indicating better understanding.
Patient reported pain related to arthritis | 3-month and 6-month intervals
  Patient reported pain related to arthritis on a visual analogue scale. The visual analogue scale is a validated measure of pain in arthritis, where participants are asked to indicate their severity of pain within the previous week on a 0 to 100mm score. A score of 0 indicates "no pain", and a score of 100 indicates "worst possible pain".

OTHER OUTCOMES:
Tender Joint Count | At the 6-month interval.
  Change in the number of tender joints as measured by their treating clinician on a 28-joint count basis.
Swollen joint count | At the 6-month interval.
  Change in the number of swollen joints as measured by their treating clinician on a 28-joint count basis.
Number of Emergency Department Visits During the Study Period | Cumulative over 6 months
  Number of Emergency Department Visits During the Study Period
Number of Days in Hospital During the Study Period | Cumulative over 6 months
  Number of Days in Hospital During the Study Period
Serious Infections | Cumulative over 6 months
  Number of Serious Infections Requiring Urgent Care or Emergency Department Visitation

CONTACTS AND LOCATIONS:
Overall Officials: Brent R Ohata, MD, Principal Investigator — University of British Columbia
Locations (1):
- Pender Community Health Centre, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No
We are working with a uniquely vulnerable population who are marginalized by extreme poverty, and feel that the risks of identification by sharing individual patient data outweigh the academic benefits in this study.

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-04-24): https://cdn.clinicaltrials.gov/large-docs/56/NCT07022756/Prot_SAP_000.pdf
  • Informed Consent Form (2025-04-24): https://cdn.clinicaltrials.gov/large-docs/56/NCT07022756/ICF_001.pdf